CLINICAL TRIAL: NCT06280872
Title: Prospective Unblinded Randomized Controlled Study Assessing the Physiologically Based Cord Clamping on Ventilation Duration in Moderate and Late Preterm
Brief Title: Physiologically Based Cord Clamping To Improve Neonatal Outcomes In Moderate And Late Preterm Newborns
Acronym: PhyCordPrem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: The Belgian Kids Fund (Unknown); Fonds IRIS-Recherche (Unknown); Ars Statistica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2023/Neonat/PhyCordPrem
Record Dates: First submitted 2024-01-11; First posted 2024-02-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Premature Birth; Respiratory Distress Syndrome in Premature Infant; Sepsis; Intraventricular Hemorrhage of Prematurity; Bronchodysplasia; Jaundice
Keywords: Moderate and late preterm newborn; Neonatal respiratory morbidity; Physiological based-cord clamping; Mother-infant bonding
MeSH Terms: conditions — Premature Birth; Sepsis; Jaundice; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological Based Cord Clamping (PBCC) (Experimental): In the intervention group, newborns will receive PBCC. The resuscitation table will be placed as close as possible to the mother's pelvis. Stabilization will start as soon as the infant is placed on the platform. The nurse will place the oximeter sensor on the right wrist, electrocardiogram electrodes on the chest of the newborn. Local resuscitation guidelines will be in respect of the Newborn Life support European Resuscitation Council 2021 guidelines. Stabilization of the newborn will be performed while the cord is intact and the cord will be clamped after respiratory stabilization will be achieved, de ﬁned as the establishment of regular spontaneous breathing, a heart rate above 100 bpm and oxygen saturation by pulse oximetry above 85% while using supplemental oxygen less than 0,4. If the infant does not reach the criteria for being stable, the maximum clamping time will be 10 min. After clamping, the platform will be withdrawn and placed next to the bed of the mother.
  Interventions: Other: Physiological Based Cord Clamping
- Differed Cord Clamping (DCC) (Active Comparator): In the control group, newborns will receive standard DCC defined as time based and performed at 60 seconds after birth, depending on the clinical condition of the infant, in accordance with the ERC guidelines 2021.Then infants will be transferred to a standard resuscitation table located in a stabilization room next to the operating room. Further treatment and intervention required for cardiopulmonary stabilization will be provided on the standard resuscitation table. Stabilization will start as soon as the infant is placed on the resuscitation table. The nurse will place the oximeter sensor on the right wrist, ECG electrodes on the chest and temperature probe on the right hypochondrium of the newborn. Local resuscitation guidelines will be in respect of the Newborn Life support European Resuscitation Council 2021 guidelines. The time to reach the stabilisation described above (a HR above 100 bpm and SpO 2 above 85% while using supplemental oxygen less than 0,4) is recorded.
  Interventions: Other: Differed Cord Clamping

INTERVENTIONS:
Other: Physiological Based Cord Clamping — see Arm Description
  Arms: Physiological Based Cord Clamping (PBCC)
Other: Differed Cord Clamping — see Arm Description
  Arms: Differed Cord Clamping (DCC)

SUMMARY:
Before birth, the baby's lungs are filled with fluid and babies do not use the lungs to breathe, as the oxygen comes from the placenta. As delivery approaches, the lungs begin to absorb the fluid. After vaginal delivery, the umbilical cord is clamped and cut after a delay that allows some of the blood in the umbilical cord and placenta to flow back into the baby. Meanwhile, as the baby breathes for the first time, the lungs fill with air and more fluid is pushed out. However, it does not always work out that way.

A baby born prematurely may have breathing problems because of extra fluid staying in the lungs related to the immaturity of the lung structure. Thus, the baby must breathe quicker and harder to get enough oxygen enter into the lungs. The newborn is separated from the mother to provide emergency respiratory support. Although the baby is usually getting better within one or two days, the treatment requires close monitoring, breathing help, and nutritional help as the baby is too tired to suck and swallow milk. Sometimes, the baby cannot recover well and show greater trouble breathing needing intensive care. This further separates the mother and her baby. A possible mean to help the baby to adapt better after a premature birth while staying close to the mother is to delay cord clamping when efficient breathing is established, either spontaneously or after receiving breathing help at birth. In this study, we intend to test this procedure in moderate or late preterm infants and see whether the technique helps the baby to better adapt after birth and to better initiate a deep bond with the mother.

DETAILED DESCRIPTION:
The successful transition from fetal to neonatal life is a major physiological challenge that requires the coordination of lung developmental processes, which culminate with the formation of a diffusible alveolar-capillary barrier, adequate pulmonary vasoreactivity, mature surfactant system, and clearance of lung fluid. During fetal life, gas exchange does not take place in fetal lungs but in the placenta. High pulmonary vascular resistance diverts blood flow to the left atrium through the foramen ovale and to the aorta via the ductus arteriosus. The placental circulation receives 30-50 % of the fetal cardiac output and is the major source of venous return to the fetal heart. Therefore, the umbilical venous return determines the preload for the left ventricle. Shortly before birth and during labor, the lungs undergo important transitional changes. The reabsorption of lung fluid within the airways is initiated during labor by adrenaline-induced activation of sodium channels. Uterine contractions during labor and the onset of inspiration after umbilical cord clamping generate a high transpulmonary pressure gradient leading to additional clearance of fluid from the airways into the surrounding tissue . Following the first breath and lung aeration, oxygen-induced vasodilation leads to a sudden rise in pulmonary blood flow and left atrial pressures, which closes the foramen ovale. Meanwhile, systemic vascular resistance increases above the level of pulmonary vascular resistance after placental removal, which reverses blood flow across the ductus arteriosus and induces ductal closure in response to high oxygen tension.

Premature birth can impact the success of adaptation to extrauterine life. Moderately preterm and late preterm births represented 4.4% of singleton live births in the Brussels area in 2020. Although they may be close to term, the loss of the last 4 to 8 weeks of gestation is vital to their physiologic and metabolic maturity. Because of their physiologic and metabolic immaturity, they have higher morbidity and mortality rates compared with term infants (gestational age 37 weeks). Although they may look similar to full-term infants, especially for the late preterm, the gap in the last few weeks of gestation is critical for physiological and metabolic maturation. Moderate and late preterm infants are at higher risk than term infants for a number of neonatal complications. This includes respiratory distress requiring non invasive or invasive ventilation, transient tachypnea of the newborn, intraventricular hemorrhage, periventricular leukomalacia, bacterial sepsis, apnoea, hypoglycemia, temperature instability, jaundice and hyperbilirubinaemia, feeding difficulties, neonatal intensive care admission, and also death. By contrast with lung's full-term newborn, lung of the preterm newborn presents an inability to adapt to extra-uterine life. Lung development at this time of gestation is in the saccular stage. Because of this immature lung structure, it results in delayed intrapulmonary fluid absorption, surfactant deficiency and inefficient gas exchange leading to respiratory morbidities such as transient tachypnea of the newborn, respiratory distress syndrome, persistent pulmonary hypertension. In addition, synchronicity and breath control is also immature and leads to apnea. These newborns exhibit a higher risk of positive pressure ventilation resuscitation at birth, admission to the neonatal intensive care unit (NICU), and severe hypoxic respiratory failure requiring mechanical ventilation in the most severe cases. In addition to increased neonatal morbidity, moderate or late preterm birth can impact mother-infant relationship. After delivery, immediate skin-to-skin contact during the first minute after birth is the natural process recommended to support mother-infant bonding and promote early onset of breastfeeding. Despite efforts made to start skin-to-skin contact as early as possible after delivery, immediate contact is practically difficult to implement related to the need for respiratory support for most of these newborns with incomplete transition to extrauterine life. In our institution, the infant is usually separated from the mother after umbilical cord clamping to provide first care by a pediatrician before returning on the mother's chest or on the father/partner's chest depending on parental wishes and maternal well-being during the operation and only if the condition of the newborn allows it. The separation between the mother and her newborn can be further extended in the case of NICU admission for various and multiple reasons related to prematurity.

The timing of umbilical cord clamping can profoundly affect the process of neonatal cardiorespiratory transition. Immediate cord clamping reduces the venous return to the heart, which transiently decreases heartbeats, cardiac output and cerebral blood flow before respiration initiates and pulmonary blood flow increases. Delayed cord clamping for longer than 60 seconds improves the transfusion of blood from the placenta to the newborn. Moreover, it can increase neonatal hemoglobin levels, improve long-term iron stores, and improve neurodevelopmental outcomes. Nevertheless, in both clinical research setting and daily practice, delayed cord clamping lasts rarely more than one minute during cesarean section. More recently, another approach, referred to as physiologically based cord clamping (PBCC), has been proposed to delay cord clamping up to 5 minutes after the onset of ventilation. PBCC allows to start lung aeration while on placental support and, therefore, promotes hemodynamic transition by increasing pulmonary blood flow and maintaining left ventricle preload. This strategy has been demonstrated efficient in preterm lambs and is feasible in very preterm infants, via the use of a purpose-designed resuscitation table that allows delayed cord clamping, maintenance of body temperature, and concomitant respiratory support where necessary. First experience has reported good parental acceptance of the procedure. Because PBCC has not been reported in moderate and late preterm infants, the present project aims to assess whether PBCC in moderate and late preterm infants would not be inferior to standard umbilical cord clamping with regards to adaptation to extrauterine life, respiratory morbidity, quality of mother-infant bonding, and maternal safety.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women followed-up in Brugmann University Hospital will be eligible to participate if:

* The delivery takes place between 32 0/7 and 36 6/7 weeks of gestation
* They carry singletons

Exclusion Criteria:

* Fetal anomalies including congenital malformations, anemia, and growth restriction with abnormal Dopplers.
* Abnormal placentation such as placenta previa.
* Signs of fetal distress necessitating an emergency cesarean section.
* Maternal health issue including severe anemia (defined as hemoglobin level < 7 g/dL), preeclampsia, and bleeding disorders.
* Maternal refusal of the use of blood products.
* General anesthesia for cesarian section.
* Planned cord blood banking.
* Total language barrier without possibility of translation

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Duration of non-invasive or invasive respiratory support. | from Birth to 28 days of life

SECONDARY OUTCOMES:
Rate of neonatal mortality | within 28 days of delivery
Rate of neonatal resuscitation | within first 10 minutes of life
  Neonatal resuscitation is defined as the use of a T-piece resuscitator for continuous airway positive pressure or intermittent positive pressure (with or without oxygen supplementation).
Rate of neonatal respiratory morbidity | from Birth to 28 days of life
  Neonatal respiratory morbidity includes respiratory distress syndrome, transient tachypnea of the newborn, air leak syndrome, and respiratory distress syndrome.
Number of admission to the NICU or special care baby unit | within first 72 hours of life
Length of hospitalization | Up to 8 weeks post delivery
Gestational age corrected at discharge | Up to 8 weeks post delivery
Changes in physiological variables during neonatal transition | Within first 10 minutes of life
  physiological variables includes the timing of the first breath/cry, measurements of parameters during the first 10 minutes of life (i.e., preductal oxygen saturation by pulse oximetry, respiratory rate, heart rate, and temperature), umbilical cord venous hemoglobin and gases, as well as Apgar scores at 1, 5, and 10 minutes.
Early neonatal parameters | within first 24 hours of life
  Early neonatal parameters includes body temperature (at 1, 2 and 3 hours of life) and body weight.
Hemoglobin level | At 48 hours of life
  in g/dl
Bilirubin level | At 48 hours of life
  in mg/dl
Occurrence of Neonatal adverse events | Within first 72hours of life
  Adverse events include hypoglycemia (glycemia <47 mg/dl), sepsis (positive blood culture), intraventricular hemorrhage, and the need for phototherapy
Biological markers of oxidative stress | immediately after cord clamping
Maternal perioperative parameters | up to 3 hours post delivery
  Maternal perioperative parameters include total surgical time, intraoperative intravenous fluid volume, intraoperative blood loss, uterotonic administration
Maternal postoperative hemoglobin level | At day 1 post delivery
  in g/dl
Number of maternal adverse events | within first 2 weeks after delivery
  Maternal adverse events include death, blood transfusion, postpartum hemorrhage, hysterectomy, admission in the Intensive Care Unit, wound seroma, and wound cellulitis
Maternal-infant bonding | At 2 weeks of life
  Parameters of mother-infant bonding include breastfeeding (Yes/No)
Maternal-infant bonding | At 2 weeks of life
  Parameters of mother-infant bonding include maternal depression measured by the Edinburgh Postnatal Depression Scale (EPDS) - score min = 0, score max = 30, higher score = worse outcome.
Maternal-infant bonding | At 2 weeks of life
  Parameters of mother-infant bonding include maternal depression measured by the Maternal Infant Bonding Scale (MIBS) - score min = 0, score max = 24, higher score = worse outcome
Rate of Maternal-infant bonding | At one month of life
  Parameters of mother-infant bonding include breastfeeding (Yes/No)
Rate of Maternal-infant bonding | At one month of life
  Parameters of mother-infant bonding include maternal depression measured by the Edinburgh Postnatal Depression Scale (EPDS) - score min = 0, score max = 30, higher score = worse outcome.
Rate of Maternal-infant bonding | At one month of life
  Parameters of mother-infant bonding include maternal depression measured the Maternal Infant Bonding Scale (MIBS) - score min = 0, score max = 24, higher score = worse outcome
Maternal-infant bonding | At 42 weeks of corrected age
  Brazelton Neonatal Behavioral Assessment Scale (NBAS) - score min = 1, score max = 6, higher score = better outcome
Parental satisfaction survey | At 42 weeks of corrected age
Child development assessment | At 6 months of corrected age
  The child development assessment is done using the Bayley scale IV - score min = 1 , score max = 19, higher score = better outcome
Success of PBCC | within first 10 minutes of life
  measured by the percentage of neonates in whom the procedure will be achieved without issue, identification of failed PBCC, and duration of stabilization with PBCC (defined as spontaneous breathing, heart rate (HR) >100 bpm, oxygen saturation by pulse oximetry (SpO2 ) ≥ 85% with inspired oxygen fraction < 0.4).

CONTACTS AND LOCATIONS:
Overall Officials: Anna AMORUSO, Principal Investigator — HUDERF
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels